CLINICAL TRIAL: NCT00605215
Title: A Multinational, Multicenter, Randomized, Parallel-Group Study Performed in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS) to Assess the Efficacy, Safety and Tolerability of Laquinimod Over Placebo in a Double-blind Design and of a Reference Arm of Interferon β-1a (Avonex®) in a Rater-blinded Design
Brief Title: BRAVO Study: Laquinimod Double-blind Placebo-controlled Study in Participants With Relapsing-Remitting Multiple Sclerosis (RRMS) With a Rater Blinded Reference Arm of Interferon β-1a (Avonex®)
Acronym: BRAVO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-LAQ-302; 2007-005450-23 (EudraCT Number)
Record Dates: First submitted 2008-01-08; First posted 2008-01-30 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — laquinimod; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 1 capsule of placebo matching to laquinimod orally once daily for 24 months.
  Interventions: Drug: Placebo
- Laquinimod (Experimental): Participants will receive 1 capsule of laquinimod 0.6 mg orally once daily for 24 months.
  Interventions: Drug: Laquinimod
- Avonex® (Active Comparator): Participants will receive an injection of Avonex® 30 micrograms (mcg) given intramuscularly (IM) once weekly for 24 months.
  Interventions: Drug: Avonex®

INTERVENTIONS:
Drug: Laquinimod — Laquinimod will be administered per dose and schedule specified in the arm description.
  Arms: Laquinimod
Drug: Placebo — Placebo matching to laquinimod will be administered per schedule specified in the arm description.
  Arms: Placebo
Drug: Avonex® — Avonex® will be administered per dose and schedule specified in the arm description.
  Other Names: Interferon β-1a
  Arms: Avonex®

SUMMARY:
The study aims to compare the effect of daily oral treatment of laquinimod capsules 0.6 milligrams (mg) with the effect of placebo capsules (capsules that contain no active medication) as well as with the effect of an existing Multiple Sclerosis (MS) injectable drug: Interferon β-1a (Avonex®).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a confirmed and documented MS diagnosis as defined by the Revised McDonald criteria [Ann Neurol 2005: 58:840-846], with a relapsing-remitting disease course.
2. Subjects must be ambulatory with converted Kurtzke EDSS score of 0-5.5.
3. Subjects must be in a stable neurological condition between screening (month -1) and baseline visits (month 0).
4. Subjects must have had experienced one of the following:
5. At least one documented relapse in the 12 months prior to screening
6. At least two documented relapses in the 24 months prior to screening
7. One documented relapse between 12 and 24 months prior to screening with at least one documented T1-Gd enhancing lesion in an MRI performed within 12 months prior to screening.
8. Subjects must be between 18 and 55 years of age, inclusive.
9. Subjects must have disease duration of at least 6 months (from first symptom) prior to screening.
10. Women of child-bearing potential must practice 2 acceptable methods of birth control [acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy or double-barrier method (condom or diaphragm with spermicide)].
11. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. An onset of relapse or any treatment with corticosteroids (intravenous [iv], intramuscular [im] and/or per os [po]) or ACTH between month -1 (screening) and 0 (baseline).
2. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
3. Use of immunosuppressive (including Mitoxantrone (Novantrone®) or cytotoxic agents within 6 months prior to the screening visit.
4. Previous use of either of the following: natalizumab (Tysabri®), cladribine or laquinimod.
5. Previous treatment with glatiramer acetate (Copaxone®) or IVIG within 3 months prior to screening visit.
6. Previous treatment with Interferon beta-1a (Avonex® or Rebif®) or Interferon beta-1b (Betaseron®).
7. Systemic corticosteroid treatment of ≥30 consecutive days duration within 2 months prior to screening visit.
8. Previous total body irradiation or total lymphoid irradiation.
9. Previous stem-cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
10. A known history of tuberculosis.
11. Acute infection 2 weeks prior to baseline visit.
12. Major trauma or surgery 2 weeks prior to baseline visit.
13. A history of vascular thrombosis (excluding catheter-site superficial venous thrombophlebitis).
14. A carrier state of factor V Leiden mutation (either homo- or heterozygous) by history or as disclosed at screening.
15. Positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or HIV antibody as disclosed at screening visit.
16. Use of potent inhibitors of CYP3A4 within 2 weeks prior to baseline visit (see detailed list of drugs in protocol) (1 month for fluoxetine).
17. Use of amiodarone within 2 years prior to screening visit.
18. Pregnancy or breastfeeding.
19. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests or chest X-ray. Such conditions may include:

    * A cardiovascular or pulmonary disorder that cannot be well-controlled by standard treatment permitted by the study protocol.
    * A gastrointestinal disorder that may affect the absorption of study medication.
    * Renal, metabolic, endocrinological or hematological diseases.
    * Any form of chronic liver disease, including known non-alcoholic steatohepatitis.
    * A ≥2xULN serum elevation of either of the following at screening: ALT, AST or direct bilirubin.
    * A QTc interval (obtained from either two ECG recordings at screening or from the mean value calculated from three measurements at baseline visit) which is ≥450msec.
    * A family history of Long-QT syndrome.
    * A history of drug and/or alcohol abuse.
    * Major psychiatric disorder.
    * A history of a convulsive disorder.
    * Known hypersensitivity to either of the following: mannitol, meglumine or sodium stearyl fumarate.
    * Known hypersensitivity that would preclude administration of laquinimod.
20. The subject's inability to give informed consent, or to complete the study, or if the subject is considered by the investigator to be, for any reason, an unsuitable candidate for this study.
21. A known history of sensitivity to Gadolinium.
22. Inability to successfully undergo MRI scanning.
23. A known history of hypersensitivity to natural or recombinant interferon beta, human albumin, or any other component of the formulation of Avonex®.
24. Subjects who suffer from any form of progressive MS
25. Any condition which the investigator feels may interfere with participation in the study
26. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation
27. Subjects who received any investigational medication, immunosuppressives or cytotoxic agents within 6 months prior to screening
28. Previous treatment with immunomodulators within two months prior to screening
29. Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1331 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2011-06-10 (Actual); Study Completion 2011-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (170):
- United States (36):
  - Teva Investigational Site 1267, Birmingham, Alabama
  - Teva Investigational Site 1237, Phoenix, Arizona
  - Teva Investigational Site 1252, Phoenix, Arizona
  - Teva Investigational Site 1279, Phoenix, Arizona
  - Teva Investigational Site 1276, Tucson, Arizona
  - Teva Investigational Site 1272, Pasadena, California
  - Teva Investigational Site 1238, Sacramento, California
  - Teva Investigational Site 1280, Aurora, Colorado
  - Teva Investigational Site 1255, Orlando, Florida
  - Teva Investigational Site 1282, Sarasota, Florida
  - Teva Investigational Site 1275, Atlanta, Georgia
  - Teva Investigational Site 1250, Peoria, Illinois
  - Teva Investigational Site 1260, Indianapolis, Indiana
  - Teva Investigational Site 1268, Lenexa, Kansas
  - Teva Investigational Site 1277, New Orleans, Louisiana
  - Teva Investigational Site 1263, Shreveport, Louisiana
  - Teva Investigational Site 1269, Baltimore, Maryland
  - Teva Investigational Site 1274, Grand Rapids, Michigan
  - Teva Investigational Site 1239, Lebanon, New Hampshire
  - Teva Investigational Site 1265, Teaneck, New Jersey
  - Teva Investigational Site 1273, Albany, New York
  - Teva Investigational Site 1264, Amherst, New York
  - Teva Investigational Site 1283, Cedarhurst, New York
  - Teva Investigational Site 1249, Raleigh, North Carolina
  - Teva Investigational Site 1262, Winston-Salem, North Carolina
  - Teva Investigational Site 1261, Akron, Ohio
  - Teva Investigational Site 1241, Canton, Ohio
  - Teva Investigational Site 1245, Cleveland, Ohio
  - Teva Investigational Site 1247, Columbus, Ohio
  - Teva Investigational Site 1244, Portland, Oregon
  - Teva Investigational Site 1258, Philadelphia, Pennsylvania
  - Teva Investigational Site 1281, Nashville, Tennessee
  - Teva Investigational Site 1284, San Antonio, Texas
  - Teva Investigational Site 1248, Richmond, Virginia
  - Teva Investigational Site 1270, Roanoke, Virginia
  - Teva Investigational Site 1253, Tacoma, Washington
- Bulgaria (17):
  - Teva Investigational Site 5914, Pleven
  - Teva Investigational Site 5915, Pleven
  - Teva Investigational Site 5917, Plovdiv
  - Teva Investigational Site 4212, Rousse
  - Teva Investigational Site 5916, Shumen
  - Teva Investigational Site 5920, Sofia
  - Teva Investigational Site 5907, Sofia
  - Teva Investigational Site 5910, Sofia
  - Teva Investigational Site 5909, Sofia
  - Teva Investigational Site 5919, Sofia
  - Teva Investigational Site 5906, Sofia
  - Teva Investigational Site 5908, Sofia
  - Teva Investigational Site 5911, Sofia
  - Teva Investigational Site 5912, Sofia
  - Teva Investigational Site 5918, Stara Zagora
  - Teva Investigational Site 5913, Varna
  - Teva Investigational Site 4211, Veliko Tarnovo
- Croatia (6):
  - Teva Investigational Site 6003, Osijek
  - Teva Investigational Site 6004, Split
  - Teva Investigational Site 6005, Varaždin
  - Teva Investigational Site 6001, Zagreb
  - Teva Investigational Site 6002, Zagreb
  - Teva Investigational Site 6006, Zagreb
- Czechia (5):
  - Teva Investigational Site 5422, Brno
  - Teva Investigational Site 5419, Olomouc
  - Teva Investigational Site 5418, Prague
  - Teva Investigational Site 5420, Praha 5- Motol
  - Teva Investigational Site 5421, Teplice
- Estonia (3):
  - Teva Investigational Site 5508, Kohtla-Järve
  - Teva Investigational Site 5507, Tallinn
  - Teva Investigational Site 5509, Tartu
- Georgia (3):
  - Teva Investigational Site 8102, Tbilisi
  - Teva Investigational Site 8104, Tbilisi
  - Teva Investigational Site 8103, Tbilisi
- Germany (8):
  - Teva Investigational Site 6701, Bayreuth
  - Teva Investigational Site 6703, Berlin
  - Teva Investigational Site 6402, Berlin
  - Teva Investigational Site 6700, Berlin
  - Teva Investigational Site 6702, Dresden
  - Teva Investigational Site 6401, Hanover
  - Teva Investigational Site 6403, Münster
  - Teva Investigational Site 6400, Ulm
- Israel (4):
  - Teva Investigational Site 8043, Haifa
  - Teva Investigational Site 8041, Jerusalem
  - Teva Investigational Site 8040, Ramat Gan
  - Teva Investigational Site 8042, Ramat Gan
- Italy (12):
  - Teva Investigational Site 3056, Bologna
  - Teva Investigational Site 3062, Catania
  - Teva Investigational Site 3053, Cefalù
  - Teva Investigational Site 3054, Chieti
  - Teva Investigational Site 3061, Empoli
  - Teva Investigational Site 3049, Florence
  - Teva Investigational Site 3055, Napoli
  - Teva Investigational Site 3048, Rome
  - Teva Investigational Site 3052, Rome
  - Teva Investigational Site 3050, Rome
  - Teva Investigational Site 3060, Rome
  - Teva Investigational Site 3051, Torino
- Lithuania (2):
  - Teva Investigational Site 5708, Kaunas
  - Teva Investigational Site 5707, Šiauliai
- North Macedonia (3):
  - Teva Investigational Site 6502, Bitola
  - Teva Investigational Site 6500, Skopje
  - Teva Investigational Site 6501, Skopje
- Poland (18):
  - Teva Investigational Site 5337, Bialystok
  - Teva Investigational Site 5329, Gdansk
  - Teva Investigational Site 5338, Gdansk
  - Teva Investigational Site 4213, Gmina Końskie
  - Teva Investigational Site 6602, Gorzów Wielkopolski
  - Teva Investigational Site 5333, Grodzisk Mazowiecki
  - Teva Investigational Site 5339, Katowice
  - Teva Investigational Site 5334, Katowice
  - Teva Investigational Site 6603, Kielce
  - Teva Investigational Site 5332, Kościerzyna
  - Teva Investigational Site 5345, Krakow
  - Teva Investigational Site 5328, Lodz
  - Teva Investigational Site 5330, Olsztyn
  - Teva Investigational Site 5331, Szczecin
  - Teva Investigational Site 5340, Warsaw
  - Teva Investigational Site 5341, Warsaw
  - Teva Investigational Site 5336, Warsaw
  - Teva Investigational Site 5335, Wroclaw
- Teva Investigational Site 1243, Guaynabo, Puerto Rico
- Romania (8):
  - Teva Investigational Site 5218, Bucharest
  - Teva Investigational Site 5214, Bucharest
  - Teva Investigational Site 5213, Bucharest
  - Teva Investigational Site 5215, Cluj-Napoca
  - Teva Investigational Site 5217, Constanța
  - Teva Investigational Site 8209, Craiova
  - Teva Investigational Site 5216, Iași
  - Teva Investigational Site 5219, Sibiu
- Russia (11):
  - Teva Investigational Site 5043, Barnaul
  - Teva Investigational Site 5033, Moscow
  - Teva Investigational Site 5032, Moscow
  - Teva Investigational Site 5041, Moscow
  - Teva Investigational Site 5038, Novosibirsk
  - Teva Investigational Site 5042, Novosibirsk
  - Teva Investigational Site 5036, Saint Petersburg
  - Teva Investigational Site 5035, Saint Petersburg
  - Teva Investigational Site 5034, Saint Petersburg
  - Teva Investigational Site 5037, Samara
  - Teva Investigational Site 5044, Ufa
- Slovakia (4):
  - Teva Investigational Site 6200, Bratislava
  - Teva Investigational Site 6201, Bratislava
  - Teva Investigational Site 6202, Nitra
  - Teva Investigational Site 6203, Žilina
- South Africa (7):
  - Teva Investigational Site 9007, Bloemfontein
  - Teva Investigational Site 9001, Cape Town
  - Teva Investigational Site 9004, Johannesburg
  - Teva Investigational Site 9003, Johannesburg
  - Teva Investigational Site 9008, Pietermaritzburg
  - Teva Investigational Site 9005, Pretoria
  - Teva Investigational Site 9006, Rosebank
- Spain (7):
  - Teva Investigational Site 3147, Barcelona
  - Teva Investigational Site 3154, Figueres-Girona
  - Teva Investigational Site 3149, L'Hospitalet de Llobregat
  - Teva Investigational Site 3152, Madrid
  - Teva Investigational Site 3151, Málaga
  - Teva Investigational Site 3148, Seville
  - Teva Investigational Site 3153, Tortosa-Tarragona
- Ukraine (15):
  - Teva Investigational Site 6503, Chernihiv
  - Teva Investigational Site 5823, Chernivtsi
  - Teva Investigational Site 5811, Dnipropetrovsk
  - Teva Investigational Site 5812, Donetsk
  - Teva Investigational Site 5814, Ivano-Frankivsk
  - Teva Investigational Site 5817, Kharkiv
  - Teva Investigational Site 5818, Kharkiv
  - Teva Investigational Site 5815, Kharkiv
  - Teva Investigational Site 5822, Kyiv
  - Teva Investigational Site 5809, Lviv
  - Teva Investigational Site 5820, Odesa
  - Teva Investigational Site 5821, Poltava
  - Teva Investigational Site 5810, Vinnytsia
  - Teva Investigational Site 5819, Zaporizhzhya
  - Teva Investigational Site 5816, Zaporizhzhya

REFERENCES:
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Kolb-Sobieraj C, Gupta S, Weinstock-Guttman B. Laquinimod therapy in multiple sclerosis: a comprehensive review. Neurol Ther. 2014 May 6;3(1):29-39. doi: 10.1007/s40120-014-0017-6. eCollection 2014 Jun. PMID 26000222

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 1 capsule of placebo matched to laquinimod orally once daily for 24 months.
- Laquinimod: Participants received 1 capsule of laquinimod 0.6 millograms (mg) orally once daily for 24 months.
- Avonex®: Participants received an injection of Avonex® 30 micrograms (mcg) given intramuscularly (IM) once weekly for 24 months.
Period: Overall Study
Arm/Group | Placebo | Laquinimod | Avonex®
Started | 450 | 434 | 447
Received at Least 1 Dose of Study Drug | 449 | 433 | 442
Completed | 359 | 353 | 378
Not Completed | 91 | 81 | 69
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 19 | 21 | 26
Not completed — Refusal to sign the re-consent form | 8 | 3 | 3
Not completed — Withdrawal by Subject | 39 | 37 | 27
Not completed — Request of Primary Care Physician or Investigator | 6 | 4 | 4
Not completed — Protocol Violation | 3 | 4 | 1
Not completed — Pregnancy | 8 | 5 | 4
Not completed — Lost to Follow-up | 8 | 5 | 2
Not completed — Other than specified | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Laquinimod: Participants received 1 capsule of laquinimod 0.6 mg orally once daily for 24 months.
- Avonex®: Participants received an injection of Avonex® 30 mcg given IM once weekly for 24 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Laquinimod | Avonex® | Total
Number analyzed (Participants) | 450 | 434 | 447 | 1331
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (9.5) | 37.0 (9.3) | 38.2 (9.5) | 37.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 321 | 282 | 307 | 910
  Male | 129 | 152 | 140 | 421
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 2
  Black of African Heritage | 1 | 1 | 0 | 2
  Black/African American | 2 | 1 | 4 | 7
  White | 443 | 426 | 440 | 1309
  Hispanic | 3 | 3 | 1 | 7
  Other | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Confirmed Relapses
Description: A relapse was defined as the appearance of new neurological abnormalities or the reappearance of previously observed neurological abnormalities; lasting at least 48 hours and immediately preceded by an improved neurological state of ≥30 days from onset of previous relapse, accompanied by observed objective neurological changes (an increase of ≥0.5 in Expanded Disability Status Scale [EDSS] score, or an increase of 1 grade in the score of 2 or more of the 7 Functional Systems [FS], or an increase of 2 grades in the score of 1 FS as compared to the previous evaluation). Total number of confirmed relapses during the treatment period was divided by the sum of number of days on study in the treatment period and then multiplied by the number of days in the year to calculate the annualized relapse rate. Annualized relapse rate was derived from a baseline-adjusted negative binomial regression.
Time Frame: Baseline up to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Mean (95% Confidence Interval); unit: relapse per year
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 450 | 434 | 447
relapse per year | 0.344 [0.291 to 0.406] | 0.283 [0.237 to 0.337] | 0.255 [0.213 to 0.304]
Statistical Analysis 1: Comparison: Placebo vs Laquinimod; Analysis was performed using baseline-adjusted negative binomial regression, where a participant's number of relapses during the double-blind, placebo-controlled phase served as the response variable and an offset based on the log of participant's exposure in years was employed to adjust for variability of treatment exposure. The model included baseline EDSS score, log of (prior 2-year number of relapses+1) and CGR as covariates; Test type: Other; p = 0.0746, Negative Binomial Regression — Threshold for significance at 0.05 level; Risk Ratio (RR) = 0.823, 95% CI 2-sided [0.664 to 1.020], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: Placebo vs Avonex®; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0067, Negative Binomial Regression; Risk Ratio (RR) = 0.741, 95% CI 2-sided [0.596 to 0.920], Standard Error of Mean 0.082

2. Secondary Outcome: Change From Baseline in Disability as Assessed by the Multiple Sclerosis Functional Composite (MSFC) Score
Description: The Multiple Sclerosis Functional Composite is an instrument assessing disability that consists of 3 clinical assessments. The 3 are Timed 25-Foot Walk, 9-Hole Peg Test which measures upper extremity (arm and hand) function, and PASAT (Paced Auditory Serial Addition Test) which is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. A Z-score is used to define a common metric from the 3 assessments that constitute the MSFC score. The study's population at baseline was used as reference population for the Z-score calculation. A Z-score of 0 represents the population mean at baseline. Higher Z-scores correspond to an improved outcome.
Time Frame: Baseline, Month 24
Population: ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 358 | 351 | 377
Z score | -0.5 (0.85) | -0.00 (0.85) | -0.01 (0.75)

3. Secondary Outcome: Percent Change From Baseline in Brain Volume
Description: Change in brain volume was derived from MRI scans obtained at baseline and at Month 24.
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 341 | 332 | 361
Percent Change | -0.53 (0.65) | -0.51 (0.65) | -0.53 (0.65)

4. Secondary Outcome: Accumulation of Physical Disability Measured by the Number of Participants With Confirmed Progression of EDSS
Description: A confirmed progression of EDSS was defined as a 1 point increase from baseline on EDSS score if baseline EDSS was between 0 and 5.0, or a 0.5 point increase if baseline EDSS was 5.5, confirmed 3 months later. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]). Data is presented as distribution of confirmed progression (number of participants with confirmed progression of EDSS) sustained for 3 months. Progression could not be confirmed during a relapse.
Time Frame: Baseline up to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 450 | 434 | 447
Participants | 60 | 42 | 47

5. Other Pre Specified Outcome: Change From Baseline in General Health Status as Assessed by the Short-Form General Health Survey (SF-36) Patient-Reported Questionnaire For Physical Component Summary (PCS) Scores
Description: The SF-36 questionnaire has 36 questions composing the scale that represent 8 domains: 1) physical functioning, role physical, 2) bodily pain, 3) general health, 4) vitality, 5) social functioning, 6) role, 7) emotional, and 8) mental health. The scores for the 8 domains were combined into two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score. Items 1 to 4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item were summed and averaged (range: 0=worst to 100=best). Higher scores represent better health status and functional ability.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 450 | 434 | 447
units on a scale
  Month 6: number analyzed (Participants) | 414 | 397 | 414
  Month 6 | -0.2 (6.3) | 0.1 (6.3) | -0.1 (6.3)
  Month 12: number analyzed (Participants) | 385 | 377 | 402
  Month 12 | -0.3 (6.9) | -0.1 (6.9) | 0.0 (6.7)
  Month 18: number analyzed (Participants) | 364 | 361 | 379
  Month 18 | -0.5 (7.0) | -0.3 (7.0) | 0.2 (6.9)
  Month 24: number analyzed (Participants) | 356 | 348 | 374
  Month 24 | -0.6 (7.6) | 0.1 (6.9) | 0.2 (7.0)

6. Other Pre Specified Outcome: Change From Baseline in General Health Status as Assessed by the Short-Form General Health Survey (SF-36) Patient-Reported Questionnaire For Mental Component Summary (MCS) Scores
Description: as for outcome 5
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 450 | 434 | 447
units on a scale
  Month 6: number analyzed (Participants) | 414 | 397 | 414
  Month 6 | -0.4 (8.5) | -0.6 (8.2) | -0.4 (8.9)
  Month 12: number analyzed (Participants) | 385 | 377 | 402
  Month 12 | -0.7 (9.2) | -0.1 (9.8) | -0.5 (9.0)
  Month 18: number analyzed (Participants) | 364 | 361 | 379
  Month 18 | -0.9 (9.3) | -1.4 (10.4) | -0.7 (9.2)
  Month 24: number analyzed (Participants) | 356 | 348 | 374
  Month 24 | -0.5 (9.2) | -0.9 (9.6) | -0.3 (9.3)

7. Other Pre Specified Outcome: Cumulative Number of New or Enlarging Hypointense Lesions on Enhanced T1 Scans
Description: The cumulative number of new or enlarging hypointense lesions was calculated as the sum of the numbers of new or enlarging hypointense lesions observed on scans taken at Months 12 and 24.
Time Frame: Months 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 393 | 381 | 403
lesions | 7.10 (10.25) | 7.33 (10.87) | 5.91 (8.58)

8. Other Pre Specified Outcome: Cumulative Number of Enhancing Lesions on T1-Weighted Images
Description: The cumulative number of T1 Gadolinium (Gd)-enhancing lesions was calculated as the sum of the numbers of Gd-enhancing lesions observed on scans taken at Months 12 and 24.
Time Frame: Months 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Laquinimod | Avonex®
Number analyzed (Participants) | 393 | 381 | 404
lesions | 2.70 (8.00) | 2.58 (7.40) | 1.23 (3.32)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: Safety analysis set included all randomized participants who received at least 1 dose of laquinimod.
Arm/Group | Placebo | Laquinimod | Avonex®
All-Cause Mortality (participants affected / at risk) | 0/449 | 1/433 | 1/442
Serious Adverse Events (participants affected / at risk) | 36/449 | 31/433 | 25/442
Other Adverse Events (participants affected / at risk) | 146/449 | 158/433 | 286/442
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=449) | Laquinimod (N=433) | Avonex® (N=442)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Measles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia measles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Myelitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Sperm granuloma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acoustic neuroma removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Internal fixation of spine (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Lymphadenectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Orchidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Radical hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal cord operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=449) | Laquinimod (N=433) | Avonex® (N=442)
Influenza like illness (General disorders) | 7 (7) | 5 (5) | 206 (385)
Pyrexia (General disorders) | 7 (10) | 6 (7) | 52 (77)
Influenza (Infections and infestations) | 28 (32) | 27 (30) | 20 (30)
Nasopharyngitis (Infections and infestations) | 35 (45) | 40 (63) | 29 (37)
Upper respiratory tract infection (Infections and infestations) | 36 (43) | 34 (41) | 22 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (26) | 24 (27) | 18 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (50) | 44 (61) | 15 (30)
Headache (Nervous system disorders) | 53 (105) | 54 (100) | 60 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.